CLINICAL TRIAL: NCT06240689
Title: A Prospective Randomized Controlled Study of Immune Checkpoint Maintenance Therapy After Radiotherapy and Chemotherapy for Locally Advanced Head And Neck Tumors Based on Peripheral Blood CD8Tex Detection in Peripheral Blood
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y2023-0889
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — sintilimab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional arm (Experimental): The experimental group started treatment within 1 month after the end of chemoradiotherapy, and Sintilimab was given intravenously on the first day of each cycle, and a cycle of 21 days, and a total of 18 cycles were expected to be administered, or until disease progression.
  Interventions: Drug: Sintilimab
- Control arm (Placebo Comparator): The control group started treatment within 1 month after the end of chemoradiotherapy, and placebo was given intravenously on the first day of each cycle, and a cycle of 21 days, and a total of 18 cycles were expected to be administered, or until disease progression.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sintilimab — Sintilimab is administered intravenously on the first day of each cycle. 21 days per cycle.
  Other Names: IBI308
  Arms: Interventional arm
Drug: Placebo — Placebo is administered intravenously on the first day of each cycle. 21 days per cycle.
  Other Names: 0.9% sodium chloride solution
  Arms: Control arm

SUMMARY:
The goal of this prospective, randomized, single-blind controlled clinical study is to explore the efficacy of maintenance therapy with Sintilimab after chemoradiotherapy in locally advanced head and neck squamous cell carcinoma. The main questions it aims to answer are:

How works well the Sintilimab was in the treatment group？ How safe the Sintilimab is？ Participants will intravenous Sintilimab or placebo (a look-alike substance that contains no active drug) within 1 month after the end of chemoradiotherapy, and 21 days is a cycle. Blood tests, electrocardiogram are rechecked every 2 cycles, and CT was rechecked every 4 cycles to evaluate toxicity and side effects and recurrence.

Researchers will compare invention group to control group to see if the Sintilimab works well.

DETAILED DESCRIPTION:
The experimental group and the control group start treatment within 1 month after the end of chemoradiotherapy, and Sintilimab was given intravenously on the first day of each cycle in the experimental group while placebo was given in the control group, and a cycle of 21 days, and a total of 18 cycles were expected to be administered, or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years old, ≤ 75 years old.
2. Histologically confirmed inoperable locally advanced head and neck tumor T3 or N+ or above.
3. Patients undergoing concurrent chemoradiotherapy
4. ECOG performance status of 0 to 1.
5. Life expectancy of at least 12 weeks.
6. At least one measurable lesion
7. Blood test: absolute neutrophil count (ANC) > 1.5×109/L, hemoglobin > 8g/dL and platelet > 100 ×109/L (subject to the normal value of the clinical trial center).
8. Prothrombin time (PT) <1.5 times the upper limit of normal and normal thromboplastin time (APTT) <1.5 times the upper limit of normal.
9. Laboratory examination, serum creatinine less than or equal to 1.5 times the upper limit of the reference range of normal values (If serum creatinine is elevated, 24-hour urine must be collected. Except for the 24-hour creatinine clearance rate is > 50ml/min).
10. In the absence of liver metastases, ALT or AST is less than or equal to 2.5 times the upper limit of the reference range of normal values, and total serum bilirubin is less than or equal to 1.5 times the upper limit of the reference range of normal values; for patients with liver metastases, ALT or AST is less than or equal to 5 times the upper limit of the reference range of normal values, and total serum bilirubin is less than or equal to 3 times of the upper limit of the reference range of normal values.
11. Females of childbearing potential must be willing to use adequate contraception for the duration of study drug treatment.
12. Signed informed consent.
13. At the end of radiotherapy, the proportion of PD1+CD8T cells in peripheral blood is greater than 10%, or more than 2 times higher than baseline

Exclusion Criteria:

1. Active autoimmune disease requiring systemic therapy (i.e., use of disease-modifying medications, corticosteroids, or immunosuppressants) within the previous 2 years. Replacement therapies (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) are not considered systemic treatments.
2. Diagnosed with immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial therapy. After consultation with the sponsor, the use of physiologic doses of corticosteroids may be approved.
3. Other malignancies that are known to be progressing or requiring active treatment. Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix that has received curative therapy are excluded.
4. Have an active infection requiring systemic therapy.
5. Medical history or evidence of disease that may confound the results of the trial, prevent the subject from participating in the study throughout the study, abnormal treatment or laboratory values, or the investigator believes that participation in the study is not in the best interest of the subject.
6. Known psychiatric or substance abuse disorder that may affect compliance with test requirements.
7. Female subjects who are pregnant or lactating, or who are expected to conceive during the planned trial period or up to 180 days after the last dose of study treatment, or male subjects whose spouse is preparing to become pregnant.
8. Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-01-25 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years
  progression-free survival
1-year PFS | 1 year
  1-year progression-free survival

SECONDARY OUTCOMES:
OS | 3 years
  Overall Survival
Safety and tolerability | 3 years
  All adverse events will be assessed by the investigator in accordance with NCI Common Terminology for Adverse Events (CTCAE) version 5.0.
EORTC Quality of Life Questionnaire Head and Neck (H&N)-35 scores | 3 years
  Assessment of quality of life of HNSCC

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT06240689/Prot_000.pdf
  • Informed Consent Form (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT06240689/ICF_001.pdf